CLINICAL TRIAL: NCT01266876
Title: A Randomized, Double-Blind, Placebo-Controlled, 12-Week Study of the Safety and Efficacy of REGN727 in Patients With Heterozygous Familial Hypercholesterolemia
Brief Title: Study of the Safety and Efficacy of REGN727/SAR236553 in Patients With HeFH Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R727-CL-1003
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Results first posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-08

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Placebo SC injection Q2W added to stable statin regimen with or without concomitant ezetimibe for 12 weeks.
  Interventions: Drug: Placebo
- Alirocumab 150 mg Q4W (Experimental): Alirocumab 150 mg SC injection Q4W added to stable statin regimen with or without concomitant ezetimibe for 12 weeks.
  Interventions: Drug: Alirocumab
- Alirocumab 200 mg Q4W (Experimental): Alirocumab 200 mg SC injection Q4W added to stable statin regimen with or without concomitant ezetimibe for 12 weeks.
  Interventions: Drug: Alirocumab
- Alirocumab 300 mg Q4W (Experimental): Alirocumab 300 mg SC injection Q4W added to stable statin regimen with or without concomitant ezetimibe for 12 weeks.
  Interventions: Drug: Alirocumab
- Alirocumab 150 mg Q2W (Experimental): Alirocumab 150 mg SC injection Q2W added to stable statin regimen with or without concomitant ezetimibe for 12 weeks.
  Interventions: Drug: Alirocumab

INTERVENTIONS:
Drug: Alirocumab — Alirocumab two SC injections in the abdomen only.
  Other Names: REGN727/SAR236553
  Arms: Alirocumab 150 mg Q2W; Alirocumab 150 mg Q4W; Alirocumab 200 mg Q4W; Alirocumab 300 mg Q4W
Drug: Placebo — Placebo two SC injections in the abdomen only.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of REGN727/SAR236553 in participants diagnosed with heterozygous familial hypercholesterolemia (heFH)

ELIGIBILITY:
Inclusion Criteria:

1. Must meet the World Health Organization criteria for heFH
2. Participants must be on a stable statin dose, with or without ezetimibe, for at least 6 weeks before screening
3. Serum LDL-C levels ≥ 100 mg/dL at screening
4. Willing to follow the NCEP ATPIII TLC diet, or an equivalent diet plan, starting at screening and continuing until the last study visit
5. A negative urine/serum pregnancy test at each screening visit and start of the study, for women of childbearing potential

Key Exclusion Criteria:

1. Participants with homozygous FH (clinically or by previous genotyping)
2. Use of a medication (other than a statin or EZE) to alter serum lipids within 42 days (6 weeks) before screening including, but not limited to:

   * Fibrates
   * Niacin (>500 mg/day)
   * Omega-3 fatty acids (>1000 mg/day of DHA/EPA)
   * Bile acid resins
3. Use of nutraceuticals or OTC medications that may alter lipid levels that are not stable for at least 6 weeks before screening and are not planned to remain constant throughout the study. Examples include:

   * Omega-3 fatty acids (≤1000 mg/day of DHA/EPA)
   * Niacin (≤500 mg/day)
   * Plant stanols, such as found in Benecol, flax seed oil, psyllium
   * Red yeast rice
4. Disorders known to influence lipid levels, such as nephrotic syndrome, significant liver disease, Cushing's disease, untreated hypothyroidism (patients on stable thyroid replacement for at least 12 weeks before the full screening visit, who are metabolically euthyroid by thyroid-stimulating hormone (TSH) testing are allowed)
5. Use of thyroid medications (except for replacement therapy which has been stable for at least 12 weeks before the full screening visit)
6. Fasting serum TG >350 mg/dL screening
7. LDL apheresis within 12 months before screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (22):
- United States (17):
  - Huntsville, Alabama
  - Mission Viejo, California
  - Newport Beach, California
  - Bridgeport, Connecticut
  - Jacksonville, Florida
  - Miami, Florida
  - Port Orange, Florida
  - Chicago, Illinois
  - Kansas City, Kansas
  - Auburn, Maine
  - Biddeford, Maine
  - St Louis, Missouri
  - Concord, New Hampshire
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Nashville, Tennessee
  - Houston, Texas
- Canada (5):
  - Winnipeg, Manitoba
  - London, Ontario
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Saint Foy, Quebec

REFERENCES:
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Defesche JC, Stefanutti C, Langslet G, Hopkins PN, Seiz W, Baccara-Dinet MT, Hamon SC, Banerjee P, Kastelein JJP. Efficacy of alirocumab in 1191 patients with a wide spectrum of mutations in genes causative for familial hypercholesterolemia. J Clin Lipidol. 2017 Nov-Dec;11(6):1338-1346.e7. doi: 10.1016/j.jacl.2017.08.016. Epub 2017 Sep 4. PMID 28964736
- [Derived] Toth PP, Hamon SC, Jones SR, Martin SS, Joshi PH, Kulkarni KR, Banerjee P, Hanotin C, Roth EM, McKenney JM. Effect of alirocumab on specific lipoprotein non-high-density lipoprotein cholesterol and subfractions as measured by the vertical auto profile method: analysis of 3 randomized trials versus placebo. Lipids Health Dis. 2016 Feb 13;15:28. doi: 10.1186/s12944-016-0197-4. PMID 26872608
- [Derived] Stein EA, Gipe D, Bergeron J, Gaudet D, Weiss R, Dufour R, Wu R, Pordy R. Effect of a monoclonal antibody to PCSK9, REGN727/SAR236553, to reduce low-density lipoprotein cholesterol in patients with heterozygous familial hypercholesterolaemia on stable statin dose with or without ezetimibe therapy: a phase 2 randomised controlled trial. Lancet. 2012 Jul 7;380(9836):29-36. doi: 10.1016/S0140-6736(12)60771-5. Epub 2012 May 26. PMID 22633824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 centers in the United States of America and Canada. Overall, 118 participants were screened between January 2011 and June 2011.
Pre-assignment Details: Randomization was stratified by concomitant use of ezetimibe (Yes/No). Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 1:1:1:1:1 ratio after confirmation of selection criteria. 77 participants were randomized.
Groups:
- Placebo: Placebo subcutaneous (SC) injection once every two weeks (Q2W) added to stable statin regimen with or without concomitant ezetimibe for 12 weeks.
- Alirocumab 150 mg Q4W: Alirocumab 150 mg SC injection once every 4 weeks (Q4W) added to stable statin regimen with or without concomitant ezetimibe for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Started | 15 | 15 | 16 | 15 | 16
Completed | 15 | 15 | 16 | 14 | 16
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W | Total
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (9.6) | 51.3 (7.7) | 52.9 (11.2) | 54.3 (9.6) | 56.3 (10.2) | 53.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 7 | 8 | 3 | 30
  Male | 9 | 9 | 9 | 7 | 13 | 47
Low Density Lipoprotein Cholesterol (LDL-C) in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C from Friedewald formula.
  mg/dL | 150.8 (34.0) | 166.7 (50.1) | 169.8 (57.0) | 139.6 (24.7) | 147.2 (32.6) | 154.9 (42.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-treatment Analysis
Description: Calculated LDL-C values were obtained using the Friedewald formula. Baseline adjusted least squares (LS) means and standard errors were estimated using an analysis of covariance (ANCOVA) model including available post-baseline data on treatment from first investigational medicinal product (IMP) injection up to 21 days after last IMP injection (on-treatment analysis). Missing Week 12 data were imputed by last observation carried forward [LOCF] method.
Time Frame: From Baseline to Week 12 (LOCF)
Population: Modified Intent-To-Treat (mITT) population included all randomized participants with one baseline and at least one post baseline on-treatment calculated LDL-C.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
percent change | -10.7 (5.0) | -28.9 (5.1) | -31.5 (4.9) | -42.5 (5.1) | -67.9 (4.9)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 150 mg Q2W; Each treatment group was compared to placebo using ANCOVA-derived contrasts. A hierarchical testing procedure was applied to ensure strong control of overall Type-I error rate at 0.05 level. Order was following: 1. Alirocumab 150 mg Q2W versus placebo 2. Alirocumab 300 mg Q4W versus placebo 3. Alirocumab 200 mg Q4W versus placebo 4. Alirocumab 150 mg Q4W versus placebo Testing continued only when high-order test was statistically significant at 5% level; Test type: Superiority or Other; p = 0.0000, ANCOVA — Threshold for significance at ≤ 0.05
Statistical Analysis 2: Comparison: Placebo vs Alirocumab 300 mg Q4W; Test type: Superiority or Other; p = 0.0000, ANCOVA — Threshold for significance at ≤ 0.05
Statistical Analysis 3: Comparison: Placebo vs Alirocumab 200 mg Q4W; Test type: Superiority or Other; p = 0.0035, ANCOVA — Threshold for significance at ≤ 0.05
Statistical Analysis 4: Comparison: Placebo vs Alirocumab 150 mg Q4W; Test type: Superiority or Other; p = 0.0113, ANCOVA — Threshold for significance at ≤ 0.05

2. Secondary Outcome: Absolute Change From Baseline in Calculated LDL-C at Week 12 - On-treatment Analysis
Description: Calculated LDL-C value was obtained from Friedewald formula. Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 12 (LOCF)
Population: mITT population included all randomized participants with one baseline and at least one on-treatment calculated LDL-C.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
mg/dL | -19.1 (7.9) | -42.2 (8.0) | -51.3 (7.7) | -66.9 (8.0) | -102.5 (7.6)

3. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 12 - On-treatment Analysis
Description: Calculated LDL-C value was obtained from Friedewald formula.
Time Frame: Week 12 (LOCF)
Population: mITT population included all randomized participants with one baseline and at least one on-treatment calculated LDL-C.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
percentage of participants | 13.3 | 26.7 | 18.8 | 66.7 | 93.8

4. Secondary Outcome: Percentage of Participants Achieving LDL-C < 70 mg/dL (1.81 mmol/L) at Week 12 - On-treatment Analysis
Description: Calculated LDL-C value was obtained from Friedewald formula.
Time Frame: Week 12 (LOCF)
Population: mITT population included all randomized participants with one baseline and at least one on-treatment calculated LDL-C.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
percentage of participants | 0.0 | 13.3 | 12.5 | 46.7 | 81.3

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 12 (LOCF)
Population: mITT population included all randomized participants with one baseline and at least one on-treatment total cholesterol value.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
percent change | -8.5 (3.8) | -18.1 (3.9) | -19.7 (3.7) | -25.7 (3.8) | -43.6 (3.7)

6. Secondary Outcome: Absolute Change From Baseline in Total Cholesterol at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 12 (LOCF)
Population: mITT population included all randomized participants with one baseline and at least one post baseline on-treatment total cholesterol value.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
mg/dL | -20.3 (9.4) | -40.3 (9.5) | -50.1 (9.2) | -61.7 (9.5) | -99.9 (9.1)

7. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint..
Time Frame: From Baseline to Week 12 (LOCF)
Population: mITT population included all randomized participants with one baseline and at least one on-treatment HDL-C value.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
percent change | 2.2 (3.7) | 7.9 (3.7) | 6.5 (3.5) | 1.00 (3.8) | 12.3 (3.6)

8. Secondary Outcome: Absolute Change From Baseline in HDL-C at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 12 (LOCF)
Population: mITT population included all randomized participants with one baseline and at least one post baseline HDL-C value.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
mg/dL | 0.4 (1.9) | 4.2 (1.9) | 3.3 (1.8) | 4.5 (2.0) | 6.0 (1.8)

9. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12 - On-treatment Analysis
Description: Since the assumptions of normal distribution and equality of variances were not verified for the lipid parameter, percent changes were expressed as median (interquartile range)
Time Frame: From Baseline to Week 12 (LOCF)
Population: mITT population included all randomized participants with one baseline and at least one post baseline on-treatment fasting triglycerides value.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
percent change | -10.6 [-28.5 to 9.5] | -16.7 [-30.1 to 21.1] | -13.2 [-30.9 to 7.4] | -4.9 [-17.0 to 10.3] | -16.2 [-30.7 to 25.1]

10. Secondary Outcome: Absolute Change From Baseline in Triglycerides at Week at 12 - On-treatment Analysis
Description: Since the assumptions of normal distribution and equality of variances were not verified for the lipid parameters, percent changes were expressed as median (interquartile range)
Time Frame: From Baseline to Week 12 (LOCF)
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
mg/dL | -11.0 [-89.5 to 7.5] | -20.0 [-37.0 to 13.0] | -13.5 [-35.3 to 9.5] | -3.5 [-33.0 to 6.0] | -14.8 [-64.5 to 34.0]

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 12
Population: mITT population included all randomized participants with one baseline and at least one post baseline on-treatment non-HDL-C value.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
percent change | -11.3 (4.7) | -26.8 (4.8) | -27.4 (4.6) | -39.0 (4.8) | -57.9 (4.6)

12. Secondary Outcome: Absolute Change From Baseline in Non-HDL-C at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 12 (LOCF)
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
mg/dL | -22.8 (8.8) | -46.0 (8.9) | -52.3 (8.6) | -70.6 (9.0) | -103.6 (8.5)

13. Secondary Outcome: Percent Change From Baseline in Apo Lipoprotein B (Apo-B) at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 12 (LOCF)
Population: mITT population included all randomized participants with one baseline and at least one post baseline on-treatment Apo-B value.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
percent change | -6.4 (4.2) | -20.9 (4.2) | -20.9 (4.0) | -28.4 (4.3) | -50.2 (4.0)

14. Secondary Outcome: Absolute Change From Baseline in Apo-B at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
mg/dL | -9.3 (5.5) | -24.3 (5.5) | -28.7 (5.3) | -34.7 (5.6) | -64.4 (5.3)

15. Secondary Outcome: Percent Change From Baseline in Apolipoprotein - A1 (Apo-A1) at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 12 (LOCF)
Population: mITT population included all randomized participants with one baseline and at least one post baseline on-treatment Apo-A1 value.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
percent change | -5.3 (3.1) | 2.4 (3.1) | 1.7 (2.9) | 5.6 (3.1) | 8.8 (2.9)

16. Secondary Outcome: Absolute Change From Baseline in Apo-A1 at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 12 (LOCF)
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
mg/dL | -9.7 (4.6) | 3.4 (4.5) | 2.8 (4.3) | 7.8 (4.6) | 11.0 (4.4)

17. Secondary Outcome: Absolute Change in the Ratio ApoB/ApoA-1 From Baseline to Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 12
Population: mITT population included all randomized participants with one baseline and at least one post baseline on-treatment Apo-B and ApoA-1 value.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
ratio | -0.03 (0.04) | -0.18 (0.04) | -0.20 (0.04) | -0.25 (0.04) | -0.49 (0.04)

18. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12 - On-treatment Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 12 (LOCF)
Population: mITT population included all randomized participants with one baseline and at least one post baseline on-treatment lipoprotein(a) value.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
percent change | -3.9 [-18.4 to 0.0] | -10.1 [-22.2 to 3.8] | -7.5 [-22.5 to 0.0] | -15.3 [-25.2 to 10.6] | -23.4 [-44.6 to -6.6]

19. Secondary Outcome: Absolute Change From Baseline in Lipoprotein(a) at Week 12 - On-treatment Analysis
Description: as for outcome 9
Time Frame: From Baseline to Week 12 (LOCF)
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 16
mg/dL | -2.0 [-7.0 to 0.0] | -1.5 [-10.0 to 1.5] | -1.8 [-5.0 to 0.0] | -8.0 [-19.0 to 5.0] | -11.5 [-26.0 to 1.8]

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 12
Description: Treatment emergent adverse events that developed during treatment emergent adverse events period (the time from the first dose of study drug to the last dose of study drug + 70 days (10 weeks) are reported.
Arm/Group | Placebo | Alirocumab 150 mg Q4W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Alirocumab 150 mg Q2W
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 0/16 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 9/15 | 12/15 | 13/16 | 13/15 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Alirocumab 150 mg Q4W (N=15) | Alirocumab 200 mg Q4W (N=16) | Alirocumab 300 mg Q4W (N=15) | Alirocumab 150 mg Q2W (N=16)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Alirocumab 150 mg Q4W (N=15) | Alirocumab 200 mg Q4W (N=16) | Alirocumab 300 mg Q4W (N=15) | Alirocumab 150 mg Q2W (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ocular icterus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 3 (3) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site dryness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 4 (6) | 4 (12) | 0 (0)
Injection site exfoliation (General disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 3 (4) | 0 (0) | 2 (3) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Injection site vesicles (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected bites (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure systolic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroxine decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary sediment present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.